CLINICAL TRIAL: NCT04217161
Title: Comparison of Dexcom G6 Continuous Glucose Monitoring System and Blood Glucose Levels in Adult Hemodialysis Patients With Diabetes
Brief Title: Dexcom G6 Continuous Glucose Monitoring in Hemodialysis
Acronym: DEXCOM-HD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, Irvine (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Connie Rhee, Assistant Professor of Medicine, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS# 2019-5585
Record Dates: First submitted 2020-01-02; First posted 2020-01-03 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Diabetes; Hemodialysis; Glucose Measurement
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dexcom G6 Continuous Glucose Monitor (Experimental)
  Interventions: Device: Dexcom G6 Continuous Glucose Monitor

INTERVENTIONS:
Device: Dexcom G6 Continuous Glucose Monitor — Eligible patients will undergo DDexcom G6 Continuous Glucose Monitor device placement

SUMMARY:
This is a pilot study enrolling adult hemodialysis patients with diabetes recruited from the University of California Irvine Medical Center (UCIMC) who will undergo simultaneous measurement of glucose levels using 1) continuous glucose monitor (CGM) measured by a Dexcom G6 device vs. 2) "gold-standard" blood glucose levels using capillary fingerstick or venous blood glucose measurements obtained on a point of care (POC) blood glucose meter. The study will assess Dexcom G6 accuracy by comparing glucose levels on the CGM device vs. blood glucose measurements in the study population.

ELIGIBILITY:
Inclusion Criteria:

* Adult hemodialysis patients age 18 years or older
* Have a comorbidity of diabetes
* Receipt of care from the inpatient University of California Irvine Medical Center nephrology consult service
* Expected hospital stay ≥48 hours
* Have the ability to directly provide informed consent for participation in the study

Exclusion Criteria:

* Critically-ill patients receiving care in the intensive care unit (ICU) or cardiac care unit (CCU)
* Moribund patients expected to die within 48 hours
* Presence of any condition deemed by PI's judgment that would seriously limit life expectancy (i.e., poor survival)
* Pregnant
* Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-12-21 (Estimated); Study Completion 2023-12-21 (Estimated)

PRIMARY OUTCOMES:
Blood glucose measurement | 3 to 5 days
  Proportion of CGM values within 20% of blood glucose levels >100 mg/dl or within 20 mg/dl of blood glucose level for levels <=100 mg/dl. (Will examine different thresholds of CGM values within a certain range of blood glucose levels, i.e., 10%, 15%, 25%.)

SECONDARY OUTCOMES:
Hypoglycemia events | 3 to 5 days
  Comparison in number of hypoglycemia events (glucose <70 mg/dl) determined by CGM or by blood glucose measurements

CONTACTS AND LOCATIONS:
Overall Officials: Connie Rhee, MD, MSc, Principal Investigator — Faculty
Locations (1):
- University of California Irvine, Orange, California, United States

REFERENCES:
- [Background] Rhee CM, Kovesdy CP, Ravel VA, Streja E, Brunelli SM, Soohoo M, Sumida K, Molnar MZ, Brent GA, Nguyen DV, Kalantar-Zadeh K. Association of Glycemic Status During Progression of Chronic Kidney Disease With Early Dialysis Mortality in Patients With Diabetes. Diabetes Care. 2017 Aug;40(8):1050-1057. doi: 10.2337/dc17-0110. Epub 2017 Jun 7. PMID 28592525
- [Background] Rhee CM, Kovesdy CP, Ravel VA, Streja E, Sim JJ, You AS, Gatwood J, Amin AN, Molnar MZ, Nguyen DV, Kalantar-Zadeh K. Glycemic Status and Mortality in Chronic Kidney Disease According to Transition Versus Nontransition to Dialysis. J Ren Nutr. 2019 Mar;29(2):82-90. doi: 10.1053/j.jrn.2018.07.003. Epub 2018 Nov 15. PMID 30448393
- [Background] Rhee CM, Kovesdy CP, You AS, Sim JJ, Soohoo M, Streja E, Molnar MZ, Amin AN, Abbott K, Nguyen DV, Kalantar-Zadeh K. Hypoglycemia-Related Hospitalizations and Mortality Among Patients With Diabetes Transitioning to Dialysis. Am J Kidney Dis. 2018 Nov;72(5):701-710. doi: 10.1053/j.ajkd.2018.04.022. Epub 2018 Jul 20. PMID 30037725
- [Background] Rhee CM, Leung AM, Kovesdy CP, Lynch KE, Brent GA, Kalantar-Zadeh K. Updates on the management of diabetes in dialysis patients. Semin Dial. 2014 Mar;27(2):135-45. doi: 10.1111/sdi.12198. PMID 24588802